CLINICAL TRIAL: NCT03200431
Title: Evaluation of the Influence of Output in Skin Covered by Newly Developed Adhesives
Brief Title: Evaluation of the Influence of Output on Skin Wearing a New Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_16
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of a new adhesive strip (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips on the skin after 24 hours. The adhesive strip is not yet part of a marketed ostomy device.
  Interventions: Other: New adhesive strip

INTERVENTIONS:
Other: New adhesive strip — This is a newly developed strip.

SUMMARY:
The purpose is to investigate the impact real output has on the peristomal skin covered by a newly developed adhesive.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than one year
4. Have intact skin on the area used in the evalua-tion
5. Has a stoma with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Actively participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 24 hours
  The trans epidermal water loss is measured on the peristomal skin using a probe. The Tran epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin due to natural evaporation. However, when the skin barrier is damaged the evaporation of water increases leading to a higher trans epidermal water loss. Thus, trans epidermal water loss is used to assess the damage to the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No